CLINICAL TRIAL: NCT05852847
Title: Low-dose Baricitinib Plus Danazol Versus Danazol for Patients With Steroid-resistant/Relapse Immune Thrombocytopenia: A Multicenter, Randomized, Open-label Phase 2 Trial
Brief Title: Low-dose Baricitinib Plus Danazol for Steroid-resistant/Relapse Immune Thrombocytopenia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University People's Hospital (Other)
Collaborators: Beijing Luhe Hospital (Other); Chinese PLA General Hospital (Other); Navy General Hospital, Beijing (Other); Beijing Hospital (Other Government); Beijing Friendship Hospital (Other); Peking University First Hospital (Other); Peking University Third Hospital (Other); China-Japan Friendship Hospital (Other); Beijing Tsinghua Changgeng Hospital (Other)
Responsible Party: Principal Investigator, Xiao Hui Zhang, Vice president of Peking Univeristy Institute of Hematology, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PKU-BAITP-01
Record Dates: First submitted 2023-05-02; First posted 2023-05-10 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Immune Thrombocytopenia
Keywords: Immune Thrombocytopenia; baricitinib
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — baricitinib; Danazol

STUDY DESIGN:
Intervention Model Description: Patients are randomly assigned at a 1:1 ratio to receive baricitinib plus danazol or danazol alone. Each group requires 108 patients (considering 20% drop-off) to achieve the superiority comparison.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low-dose baricitinib plus danazol (Experimental): Oral baricitinib is given at a dose of 2 mg daily for 6 months. Danazol is given at a dose of 200 mg twice a day for 6 months. Treatment will be discontinued if very severe or life-threatening adverse events developed or at the patients' request.
  Interventions: Drug: Baricitinib 2 MG [Olumiant]; Drug: Danazol
- Danazol (Active Comparator): Danazol is given at a dose of 200 mg twice a day for 6 months. Treatment will be discontinued if very severe or life-threatening adverse events developed or at the patients' request.
  Interventions: Drug: Danazol

INTERVENTIONS:
Drug: Baricitinib 2 MG [Olumiant] — Oral baricitinib was given at a dose of 2 mg daily for 6 months. Treatment was discontinued if very severe or life-threatening adverse events developed or at the patients' request.
  Other Names: Olumiant
  Arms: Low-dose baricitinib plus danazol
Drug: Danazol — Danazol was given at a dose of 200 mg bid for 6 months

SUMMARY:
This is a prospective, multicenter, randomized, controlled phase 2 trial to compare the efficacy and safety profiles in ITP patients receiving baricitinib plus danazol to those receiving danazol alone.

DETAILED DESCRIPTION:
This is a prospective, multicenter, randomized, controlled design of 216 adult patients with steroid-resistant/relapse ITP in China. Patients are randomly assigned at a 1:1 ratio to receive baricitinib plus danazol or danazol alone. Patients in the combination therapy group receive oral baricitinib at a dose of 2 mg daily and oral danazol at a dose of 200 mg twice a day. Those in the monotherapy group receive oral danazol at 200 mg twice daily. The treatment lasts for 6 months. Treatment will be discontinued if very severe or life-threatening adverse events developed or at the patients' request. The primary endpoint is durable response, defined as the maintenance of platelet count ≥ 30,000/μL, at least 2-fold increase of the baseline count, the absence of bleeding, and no need for rescue medication at the 6-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Primary immune thrombocytopenia (ITP) confirmed by excluding other supervened causes of thrombocytopenia;
2. Patients with chronic low platelet count (<30,000/μL) for 6 months who have failed at least one treatment for chronic low platelet count;
3. Patients who did not achieve a sustained response to treatment with full-dose corticosteroids for a minimum duration of 4 weeks or who relapsed during steroid-tapering or after its discontinuation;
4. Patients with a platelet count <30,000/μL or a platelet count <50,000/μL with clinically significant bleeding symptoms at the enrollment;
5. Willing and able to provide written informed consent, and agreeable to the schedule of assessment.

Exclusion Criteria:

1. Secondary immune thrombocytopenia (e.g. patients with HIV, HCV, Helicobacter pylori infection or patients with confirmed autoimmune disease);
2. Active or a history of malignancy;
3. Pregnancy or lactation;
4. Current or recent (<4 weeks prior to screening) clinically serious viral, bacterial, fungal, or parasitic infection;
5. A history of symptomatic herpes zoster infection within 12 weeks prior to screening;
6. Active or chronic viral infection from hepatitis B virus (HBV), hepatitis C virus (HCV), or human immunodeficiency virus (HIV);
7. Have evidence of active tuberculosis (TB), or have previously had evidence of active TB and did not receive appropriate and documented treatment, or have had household contact with a person with active TB and did not receive appropriate and documented prophylaxis for TB;
8. Have experienced a clinically significant thrombotic event within 24 weeks of screening or are on anticoagulants and in the opinion of the investigator are not well controlled;
9. Myocardial infarction (MI), unstable ischemic heart disease, stroke, or New York Heart Association Stage IV heart failure;
10. A history or presence of cardiovascular, respiratory, hepatic, gastrointestinal, endocrine, neurological, or neuropsychiatric disorders or any other serious and/or unstable illness that, in the opinion of the investigator, could constitute an unacceptable risk when taking investigational product or interfere with the interpretation of data;
11. Any of the following specific abnormalities on screening laboratory tests:

1) ALT or AST >2 x ULN, or total bilirubin ≥1.5 x ULN 2) hemoglobin <9 g/dL, or total white blood cell (WBC) count <2,500/µL, or neutropenia (absolute neutrophil count <1,200/µL), or lymphopenia (lymphocyte count <750/µL) 3) eGFR <50 mL/min/1.73 m^2.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2023-05-16 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Durable response | 6 months
  The maintenance of a platelet count ≥30,000/μL, at least 2-fold increase of the baseline count, the absence of bleeding, and no need for rescue medication at the 6-month follow-up.

SECONDARY OUTCOMES:
Complete response (CR) | 1 month
  A platelet count over 100,000/μL and absence of bleeding.
Response (R) | 1 month
  A platelet count over 30,000/μL and at least 2-fold increase of the baseline count and absence of bleeding.
Time to response | 6 months
  The time from starting treatment to time of achievement of CR or R.
Initial response | 28 days
  Achievement of CR or R at day 28
Bleeding events | 6 months
  Clinically significant bleeding as assessed using the world health organization (WHO) bleeding scale.
Health-related quality of life (HRQoL) | 6 months
  ITP-PAQ is used to assess the Health Related Quality of Life (HRQoL) before and after treatment.
Adverse events | 6 months
  Adverse events (AEs) are reported and graded in accordance with the Common Terminology Criteria for Adverse Events (CTCAE), version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaohui Zhang, MD, Principal Investigator — Peking University Institute of Hematology, Peking University People's Hospital
Locations (10):
- China (10):
  - Peking University Insititute of Hematology, Peking University People's Hospital, Beijing, Beijing Municipality
  - Beijing Friendship Hospital, Beijing
  - Beijing Hospital, Beijing
  - Beijing Luhe Hospital, Beijing
  - Beijing Tsinghua Changgeng Hospital, Beijing
  - China-Japan Friendship Hospital, Beijing
  - Chinese PLA General Hospital, Beijing
  - Peking University First Hospital, Beijing
  - Peking University Third Hospital, Beijing
  - The Sixth Medical Center of PLA General Hospital, Beijing